CLINICAL TRIAL: NCT01289171
Title: Acquired Epidermodysplasia Verruciformis (EV) Syndrome in HIV-infected Pediatric Patients: Prospective Treatment Trial With Topical Glycolic Acid and HPV Genotype Characterization
Brief Title: Acquired Epidermodysplasia Verruciformis (EV) Syndrome in HIV-infected Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: NeoStrata Company, Inc. (Industry); Penn Center for AIDS Research (CFAR) (Unknown)
Responsible Party: Principal Investigator, Carrie Kovarik, Professor of Dermatology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P30AI045008 (NIH)
Record Dates: First submitted 2011-01-12; First posted 2011-02-03 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Flat Warts; HIV
Keywords: The efficacy, tolerability and safety of 15% glycolic acid lotion for treatment of diffuse flat warts among HIV+ children were investigated
MeSH Terms: interventions — glycolic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glycolic acid (Experimental): All who met the study criteria commenced once daily use of 15% glycolic acid lotion.
  Interventions: Drug: Glycolic acid

INTERVENTIONS:
Drug: Glycolic acid — Those who met the study criteria commenced once daily use of 15% glycolic acid lotion to the face and/or dorsal hands, with an increase to twice daily application as tolerated after two weeks of use.
  Other Names: Neostrata 15% Glycolic acid

SUMMARY:
Many human immunodeficiency virus (HIV)-positive children are afflicted with diffuse flat warts that have been recalcitrant to multiple treatments.The aim of this prospective study was to evaluate the efficacy, safety and tolerability of 15% glycolic acid lotion (NeoStrata) for treatment of flat warts in HIV-positive children in Botswana. Additionally, the investigators characterized the flat warts in this population, including Human Papillomavirus (HPV) type(s) and degree of immunosuppression within the patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female HIV-positive patients 7 years of age or older with at least 15 flat warts, diagnosed clinically by one dermatologist (RLM), on the face and/or dorsal hands were included in the study.

Exclusion Criteria:

* Key exclusion criteria included current use of potential wart treatments or other topical OTC products on the affected area(s).

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy of 15% glycolic acid lotion for flat warts | Patients were evaluated every two weeks for eight weeks and monthly for the next eight weeks, for a total monitoring period of 16 weeks.
  Our primary objective is to determine the efficacy of 15% glycolic acid lotion for improving the cosmetic appearance of flat warts in HIV infected children and young adults on antiretroviral therapy.
Safety and tolerability of 15% glycolic acid lotion for flat warts | Patients were evaluated every two weeks for eight weeks and monthly for the next eight weeks, for a total monitoring period of 16 weeks.
  Patients were evaluated for possible side effects of the topical medication, including erythema, scaling, burning, and irritation of the skin in the area applied.

SECONDARY OUTCOMES:
HPV typing in EV-like flat warts | Biopsies were taken at the first visit, and the HPV typing was performed on all samples after the 16 week monitoring period was complete.
  Characterize the HPV types in the flat warts in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana